CLINICAL TRIAL: NCT03115658
Title: Physical Activity and First Degree Female Relatives of Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2050-09
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Female; First-degree Relative With Breast Cancer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Participants met with a PhD level psychologist experienced with health behavior change, to set a personalized exercise goal and plan. Participants were told the studies' goal to engage in 150 minutes of moderate intensity or greater physical activity each week, based on the ACSM recommendations, but participants were allowed to set any personal goal. Participants were also instructed on how to self-monitor their physical activity.
  After the initial meeting all other intervention components were sent through the mail. The intervention consists of three types of print material that were mailed: stage-matched manuals, tailored feedback report, and tip sheets.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 12 week print based intervention

SUMMARY:
The purpose of this study is to learn more about encouraging physical activity among first degree female relatives of women with breast cancer. Physical activity can decrease a woman's risk of developing breast cancer, on average, by 20%; however, physical activity interventions have not been developed specifically for first degree female relatives of cancer patients, so currently, it is unknown whether standard physical activity interventions are sufficient for these women or if first degree female relatives would benefit from an enhanced physical activity intervention that addresses information about breast cancer risk reduction. To obtain information about first degree female relatives preferences for a physical activity intervention, this study seeks to have first degree female relatives of breast cancer patients enroll in a standard physical activity intervention developed for healthy men and women. After completion of the three month intervention, the women will be asked to participate in two, one-hour long focus group with 5-7 other participants. The first focus group is to discuss aspects of the physical activity intervention that they liked and did not like, as well as things they think may have enhanced the intervention and made it more relevant to other first-degree relative of breast cancer patients. In the second focus group, participants will be shown enhancements that were developed based on information gathered from the first focus group. Participants will be asked for their feedback on the newly developed enhancements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* Have a mother, sister, or daughter who was diagnosed with breast cancer
* Have not been diagnosed with any type of cancer except basal cell carcinoma
* Able to speak and read English
* Sedentary, defined as engaging in less than 90 minutes of moderate-intensity physical activity each week

Exclusion Criteria:

* Current of planned pregnancy for next 3 months
* Presence of a known medical condition that would make physical activity unsafe
* History of a severe psychiatric illness
* Plans to move from the area in the next 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2011-01-28 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate to vigorous physical activity | baseline to 12 weeks
  7-Day Physical Activity Recall

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hartman SJ, Dunsiger SI, Marcus BH. A pilot study of a physical activity intervention targeted towards women at increased risk for breast cancer. Psychooncology. 2013 Feb;22(2):381-7. doi: 10.1002/pon.2101. Epub 2011 Dec 2. PMID 22135183
- [Derived] Hartman SJ, Rosen RK. Breast cancer relatives' physical activity intervention needs and preferences: qualitative results. BMC Womens Health. 2017 May 19;17(1):36. doi: 10.1186/s12905-017-0392-0. PMID 28526031